CLINICAL TRIAL: NCT07376421
Title: Clinical Investigation Exploring a Newly Developed Ostomy Baseplate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP383
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device (Experimental): 4 weeks treatment with investigational device
  Interventions: Device: Incestigational device
- Comparator (Active Comparator): 4 weeks treatment with investigational device
  Interventions: Device: Comparator

INTERVENTIONS:
Device: Incestigational device — 4 weeks treatment with investigational device
  Arms: Investigational device
Device: Comparator — 4 weeks treatment with comparator
  Arms: Comparator

SUMMARY:
Peristomal skin complications (PSCs) are the predominant complication for people living with a stoma, which affect their quality of life negatively.

Among the main reasons for developing PSCs are that the peristomal skin is exposed to stomal output either due to leakage of output under the baseplate and/or imperfect cutting of the hole in the baseplate, and incorrect application creating a gap between the hole in the baseplate and the stoma.

To seal this gap, Coloplast has developed a new ostomy baseplate and the aim of the investigation is to explore the investigational device 's ability to help protect the peristomal skin.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent
* Is at least 18 years of age
* Has full legal capacity
* Has an ileostomy with consistent liquid fecal output (6-7 Bristol scale).
* Has used flat 1- or 2-piece SenSura Mio, SenSura or Assura Coloplast products for at least 14 days prior to inclusion.
* Has had the stoma for at least 90 days.
* Has a stoma size less than 40mm in diameter
* Has experienced leakage under the baseplate at least three times within the last 14 days.
* Leakage defined as output/seeping under the baseplate (see Appendix A)
* Has experienced symptoms of peristomal skin complications such as itching, burning, or pain in the peristomal area within the last 14 days.
* Has suitable peristomal skin area (assessed by investigator)
* Is able to handle the electronic diary (questionnaire/photo) themselves. If needed, a trained spouse or caretaker is allowed to assist.
* Is able to handle (apply, remove, etc.) the investigational devices themselves.
* Understands that any supporting products under the baseplate are not permissible during the investigation (except for adhesive removers) and is willing to not use these during the investigation.
* Is willing and suitable (determined by the Principal Investigator or designee) to use a flat 2-piece device during the investigation.
* Is willing to change the baseplate at least every third/fourth day during the investigation.

Exclusion Criteria:

* Is currently receiving or have within the past 60 days received radio-and/or chemotherapy.
* Low doses radio- and/or chemotherapy (assessed by Principal Investigator) is allowed for other indications than cancer.
* Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g., lotion or spray treatment.
* Is breastfeeding.
* Is pregnant based on urine pregnancy test.
* Has known hypersensitivity towards any of the investigational devices used in the investigation.
* Has a complicated stoma at baseline, as assessed by investigator (e.g., dehiscence/prolapse/hernia).
* Participates in other clinical investigations. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and is otherwise complying with the inclusion and exclusion criteria of this protocol.
* Daily use of analgesics, antihistamine or steroid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-24 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum itching scale 0-10) | 8 weeks
  Itching score (weekly max at steady state* scale 0-10).
  * To account for a possible carry-over effect, the steady state period of the treatment period begins after two weeks of investigational device or comparator use. It is anticipated that the skin will have adapted to the new device after two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark